CLINICAL TRIAL: NCT03835130
Title: Interest of Pleuropulmonary Echography Versus Standard Chest X-ray in the Post-operative Follow-up of Pleuropulmonary Surgery
Brief Title: Pleuropulmonary Echography Versus Standard Chest X-ray in the Post-operative Follow-up of Pleuropulmonary Surgery
Acronym: REC
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 18_RIPH3-06
Record Dates: First submitted 2018-10-30; First posted 2019-02-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Pleuro-pulmonary Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In postoperative pleuro-pulmonary surgery, the monitoring of the appearance of complications is guided, depending on the centres, by the systematic daily performance or, in the event of a call point, by chest x-ray at the patient's bed until the drains are ablative.

This repeated performance of radiographs results in irradiation of patients but also of medical staff and a significant cost.

In the thoracic study, ultrasound imaging is a fast, cost-effective, non-irradiating solution that can be performed at the patient's bedside. It could guide the performance of chest x-ray, limit their number, with increased clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a higher age to 18 and undergoing pleuro-pulmonary surgery
* Hospitalized patient at Martinique University Hospital
* Patient receiving social security
* Patient giving his free and informed consent orally

Exclusion Criteria:

* Patient minor
* Woman who is pregnant and breast feeding
* Patient no giving his free and informed consent orally

Min Age: 18 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing pleuro-pulmonary surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Number of pleural disorders identified by each imaging technique | between 2 and 10 days
  Number

SECONDARY OUTCOMES:
Number of ultrasounds performed/number of chest x-ray performed | one year
  Ratio
Proportion of "negative" ultrasounds | one year
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas VENISSAC, MD-PhD, Principal Investigator — CHU de Martinique
Locations (1):
- CHU Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: Undecided